CLINICAL TRIAL: NCT03691194
Title: The Effects of 8 oz Fresh vs. Commercial Orange Juice on Blood Pressure In Normotensive Males Aged 18-59
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Cory Gheen, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 5180291
Record Dates: First submitted 2018-09-24; First posted 2018-10-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fresh orange juice (Experimental): Subject will take 8 ounces of fresh orange every day for 28 days.
  Interventions: Dietary Supplement: fresh orange juice
- concentrated orange juice (Active Comparator): Subject will take 8 ounces of concentrated orange juice every day for 28 days.
  Interventions: Dietary Supplement: concentrated orange juice

INTERVENTIONS:
Dietary Supplement: fresh orange juice — The fresh oranges will be bought from Sysco. They will be squeezed at the kitchen of School of Allied Health Professional with a juicer. They will either be squeezed the night before or on the same day. The juice will not be treated with additional preservatives or sugar. The brand of the juicer is Kitchen Aid. Eight ounces of fresh orange juice needs approximately two and half oranges. They will be put into 32 oz water bottles that were bought from Sysco, and then store them in the refrigerator. They will be given to the subjects every three or four days.
  Arms: fresh orange juice
Dietary Supplement: concentrated orange juice — The concentrated orange juice will be bought from Sysco then reconstituted. One part of concentrated orange juice needs four parts of water to reconstitute. Then, it will be measured and the reconstituted orange juice will be put into 32 oz water bottles that we bought from Sysco. They will be stored in the refrigerator. The subjects will need to get the reconstituted orange juice every three or four days.
  Arms: concentrated orange juice

SUMMARY:
The purpose of this graduate student research study is to determine the effects of drinking eight ounces of fresh vs. commercial orange juice on blood pressure in males with normal blood pressure.

DETAILED DESCRIPTION:
Visit 1

-

Beginning of the first four weeks:

Upon arrival, subjects will be given a consent form to sign. The student investigators will go over the layoutof the research study such as the procedures, and compliance with them. Then, subjects will be asked if they agree with drinking orange juice daily for two months. If they agree, they will be asked to relax for five minutes, and the student investigators will take their blood pressure reading three times using a blood pressure monitor. The subjects will complete the Perceived Stress Scale (PSS) survey before leaving. The subject will drink orange juice for 28 days.

•

Visits 2, 3, and 4:

Subjects will meet with the student investigators at a convenient location. Subjects will be asked to rest for five minutes. Student investigators will then take their blood pressure reading three times using a blood pressure monitor. The subjects will complete the PSS survey before leaving.

•

Between visit 2 and 3:

There is a washout period of approximately eight weeks. • During the first and second set of the 4

-week intervention phase, subjects will visit student investigators to retrieve orange juice samples every 3 or 4 days.

ELIGIBILITY:
Inclusion Criteria: Healthy 18-59 years old males, willing to keep the same lifestyle, not taking any medications or antioxidant supplements to control blood pressure, and do not drink any types of orange juice within 30 days.

Exclusion Criteria: Diabetic, smoke cigarettes, marijuana or electronic cigarettes, drink alcohol more than one a week, allergic to oranges, and diagnosed as hypotensive or hypertensive.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
blood pressure | change from baseline to 4 weeks
  Three readings will be taken each time and average them. If the subject's blood pressure is considered too high or low at any of the visits, they will be dropped from the study and we will suggest to them to see their primary physician.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | change from baseline to 4 weeks
  The PSS was developed by Sheldon Cohen and his colleagues, and was published in 1983. The PSS is a widely used psychological instrument to measures the level of stress. It has been used in many studies related to stress. The survey takes approximately three minutes to complete. The score ranges from 0-40. A score of 0-13 is considered low stress, 14-26 is moderate stress, and 27-40 is high stress.

CONTACTS AND LOCATIONS:
Overall Officials: Cory Gheen, MS RD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States